CLINICAL TRIAL: NCT01161446
Title: Comparisons of Public Health Screening Methods for Acute and Early HIV Infection: Home Self-Testing for HIV Infection
Brief Title: Home Self-Testing for HIV to Increase HIV Testing Frequency in Men Who Have Sex With Men (The iTest Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Public Health - Seattle and King County (Other Government); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Joanne Stekler, Assistant Professor, Division of Allergy & Infectious Diseases, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 36706; R01MH086360 (NIH); NIMH86360-1
Record Dates: First submitted 2010-07-09; First posted 2010-07-13 (Estimated); Results first posted 2017-06-07 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-05

CONDITIONS: HIV
Keywords: HIV; Home testing; Self-testing; HIV Infections/diagnosis; HIV Infections/prevention and control; AIDS Serodiagnosis; Oral fluids; Homosexuality, Male; Sexually transmitted diseases; Sexual behavior
MeSH Terms: conditions — HIV Infections; Disease; Homosexuality, Male; Sexually Transmitted Diseases; Sexual Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Home Testing (Experimental)
  Interventions: Behavioral: Home HIV self-testing with OraQuick ADVANCE® Rapid HIV-1/2 Antibody Test; Device: Home HIV self-testing with OraQuick ADVANCE® Rapid HIV-1/2 Antibody Test
- Standard Testing (No Intervention)

INTERVENTIONS:
Behavioral: Home HIV self-testing with OraQuick ADVANCE® Rapid HIV-1/2 Antibody Test — Participants in this arm will be given access to home HIV self-testing kits with the OraQuick ADVANCE® Rapid HIV-1/2 Antibody Test for use with oral fluids. They will be trained to use this device to test themselves for HIV and be able to request up to one self-testing kit per month throughout follow-up.
  Arms: Home Testing
Device: Home HIV self-testing with OraQuick ADVANCE® Rapid HIV-1/2 Antibody Test — The device is the home HIV self-testing kit that includes the OraQuick ADVANCE® Rapid HIV-1/2 Antibody Test for use on oral fluids. The kit itself is not the focus of this trial. As described in the Behavioral Intervention section, the intervention is having access to home self-testing for HIV.
  Arms: Home Testing

SUMMARY:
The purpose of this study is to determine whether the availability of home self-testing for HIV will increase HIV testing frequency among men who have sex with men without negatively impacting their risk for HIV acquisition.

DETAILED DESCRIPTION:
HIV counseling and testing remains one of the most effective HIV prevention interventions because many individuals newly diagnosed with HIV infection will alter their behaviors to reduce the risk of HIV transmission to others. In the U.S., men who have sex with men (MSM) represent the group with the greatest risk for HIV acquisition despite a high penetrance of testing, in part because their frequent exposures and infrequent testing can result in long intervals between HIV acquisition and diagnosis. Efforts to prevent HIV transmission among MSM must therefore increase the frequency of HIV testing and thereby decrease the time interval that infected individuals are unaware of their status and their potential for transmission. Home self-testing for HIV may increase the frequency of HIV testing, but there are concerns that it may also have negative consequences, including decreased access to risk reduction counseling.

We will randomize 246 MSM at high risk of HIV acquisition either to have access to home self-testing for HIV using the OraQuick ADVANCE® Rapid HIV-1/2 Antibody Test or to standard, clinic-based HIV testing for 15 months to determine the effects of home self-testing availability on HIV testing frequency and markers of risk for HIV acquisition and to assess the acceptability and ease of use of home self-testing. After screening to determine eligibility, study visits will occur at baseline and at 15 months. Both visits will include HIV/STD screening and surveys regarding HIV testing and risk behaviors. During follow-up, participants will be asked to complete brief online surveys after testing for HIV.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age ≥18
* Has sex with men
* HIV-negative
* Meets PHSKC HIV/STD Program definition of "high risk"
* Plans to live in Seattle for the next 15 months

Exclusion Criteria:

* Unable to safely and confidentially receive or store a home testing kit

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2010-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne D Stekler, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- Public Health - Seattle & King County STD Clinic, located at Harborview Medical Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Katz DA, Golden MR, Hughes JP, Farquhar C, Stekler JD. HIV Self-Testing Increases HIV Testing Frequency in High-Risk Men Who Have Sex With Men: A Randomized Controlled Trial. J Acquir Immune Defic Syndr. 2018 Aug 15;78(5):505-512. doi: 10.1097/QAI.0000000000001709. PMID 29697595

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Testing: HIV testing as usual.
Period: Overall Study
Arm/Group | Home Testing | Standard Testing
Started | 116 | 114
Completed | 98 | 99
Not Completed | 18 | 15
Not completed — Lost to Follow-up | 18 | 14
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Home Testing | Standard Testing | Total
Number analyzed (Participants) | 116 | 114 | 230
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 35.5 [27 to 45.5] | 37.5 [29 to 47] | 36 [28 to 46]
Sex: Female, Male [Count of Participants; unit: Participants] — Sex at birth
  Participants
    Female | 0 | 0 | 0
    Male | 116 | 114 | 230
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 13 | 34
  Not Hispanic or Latino | 93 | 99 | 192
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 7 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 10 | 21
  White | 90 | 79 | 169
  More than one race | 7 | 11 | 18
  Unknown or Not Reported | 3 | 7 | 10
Region of Enrollment [Number; unit: participants]
  United States | 116 | 114 | 230
Education [Count of Participants; unit: Participants]
  High school or less | 14 | 14 | 28
  Some college, Associate's, or technical training | 44 | 32 | 76
  Bachelor's degree or more | 57 | 65 | 122
  Unknown or not reported | 1 | 3 | 4
Living Situation [Count of Participants; unit: Participants]
  Alone in a house or apartment | 40 | 47 | 87
  With a sex partner, lover, or spouse | 16 | 18 | 34
  With friends or roommates | 46 | 31 | 77
  With parents, guardians, or other relatives | 4 | 12 | 16
  In school or university dormitories | 1 | 0 | 1
  No regular place to stay, couch surfing, homeless | 8 | 5 | 13
  Unknown or not reported | 1 | 1 | 2
Number of HIV tests in last year [Median (Inter-Quartile Range); unit: HIV tests] | 2 [1 to 3] | 2.5 [1 to 4] | 2 [1 to 4]
Currently tests for HIV on regular basis [Count of Participants; unit: Participants]
  Yes | 66 | 73 | 139
  No | 50 | 39 | 89
  Unknown or not reported | 0 | 2 | 2
Ever used a home HIV test [Count of Participants; unit: Participants]
  Yes | 2 | 10 | 12
  No | 113 | 104 | 217
  Unknown or not reported | 1 | 0 | 1
Gender of sex partners in last 3 months [Count of Participants; unit: Participants]
  Men | 107 | 107 | 214
  Women | 1 | 0 | 1
  Both men and women | 8 | 6 | 14
  Unknown or not reported | 0 | 1 | 1
Number of male sex partners in last 3 months [Median (Inter-Quartile Range); unit: partners] | 5 [3 to 10] | 5.5 [3 to 10] | 5 [3 to 10]
Number of male condomless anal intercourse partners in last 3 months [Median (Inter-Quartile Range); unit: partners] | 1 [0.5 to 2] | 1 [1 to 3] | 1 [1 to 3]
Any condomless anal intercourse with an HIV-discordant partner in last 3 months [Count of Participants; unit: Participants]
  Yes | 37 | 34 | 71
  No | 70 | 74 | 144
  Unknown or not reported | 9 | 6 | 15
Methamphetamine use in last 3 months [Count of Participants; unit: Participants]
  Yes | 12 | 10 | 22
  No | 103 | 103 | 206
  Unknown or not reported | 1 | 1 | 2
Inhaled nitrite use in last 3 months [Count of Participants; unit: Participants]
  Yes | 39 | 35 | 74
  No | 77 | 79 | 156
Diagnosis of bacterial sexually transmitted infection at enrollment visit [Count of Participants; unit: Participants]
  Yes | 9 | 19 | 28
  No | 107 | 95 | 202

OUTCOME MEASURES:

1. Primary Outcome: HIV Testing Frequency
Description: Number of HIV tests during follow-up reported by participants at end-of-study visit
Time Frame: 15 months
Measure: Mean (95% Confidence Interval); unit: HIV tests
Arm/Group | Home Testing | Standard Testing
Number analyzed (Participants) | 98 | 99
HIV tests | 5.3 [4.7 to 6.0] | 3.6 [3.2 to 4.0]
Statistical Analysis 1: Comparison: Home Testing vs Standard Testing; Test type: Superiority; p < 0.0001, t-test, 2 sided

2. Secondary Outcome: Condomless Anal Intercourse With HIV-positive or Unknown Status Partner in Last 3 Months
Time Frame: From 6 to 9 months and 12 to 15 months of follow-up
Population: Included "Overall Number of Participants Analyzed" as number who completed follow-up. However, only participants who responded to the question regarding non-concordant condomless anal intercourse in the last 3 months were included in this analysis for each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Home Testing | Standard Testing
Number analyzed (Participants) | 98 | 99
Participants
  Measured at 9 months: number analyzed (Participants) | 77 | 79
  Measured at 9 months | 16 | 17
  Measured at end of study (15 months): number analyzed (Participants) | 90 | 94
  Measured at end of study (15 months) | 26 | 23
Statistical Analysis 1: Comparison: Home Testing vs Standard Testing; Test type: Non-Inferiority — Non-inferiority bound: Self-testing was to be considered non-inferior to standard testing if the upper bound of the 95% confidence interval for the odds ratio fell below 2; Regression, Logistic; Used generalized estimating equations with exchangeable working correlation and robust standard errors to account for repeated measures; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.61 to 1.90] — The home testing arm represents the numerator and the standard testing arm the denominator

3. Secondary Outcome: Bacterial Sexually Transmitted Infections
Description: Includes syphilis, gonorrhea, and chlamydial infection
Time Frame: Assessed at 15 months
Population: Includes only participants who received screening for sexually transmitted infections at the end-of-study visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Home Testing | Standard Testing
Number analyzed (Participants) | 93 | 90
Participants | 5 | 11
Statistical Analysis 1: Comparison: Home Testing vs Standard Testing; Test type: Non-Inferiority — Home testing was to be considered non-inferior to standard testing with respect to STI prevalence if the upper bound of the 95% confidence interval for the difference between the two arms (home - standard) fell below 10%; Difference in proportions = -0.068, 95% CI 2-sided [-0.16 to 0.016]

4. Secondary Outcome: Number of Male Condomless Anal Intercourse Partners in Last 3 Months
Time Frame: From 6 to 9 and 12 to 15 months
Population: Included "Overall Number of Participants Analyzed" as number who completed follow-up. However, only participants who responded to the question regarding condomless anal intercourse partners in the last 3 months were included in this analysis for each time point.
Measure: Mean (Standard Error); unit: number of partners
Arm/Group | Home Testing | Standard Testing
Number analyzed (Participants) | 98 | 99
number of partners
  Measured at 9 months: number analyzed (Participants) | 80 | 80
  Measured at 9 months | 1.375 (0.207) | 2.050 (0.313)
  Measured at end of study (15 months) | 2.337 (0.355) | 2.141 (0.314)
Statistical Analysis 1: Comparison: Home Testing vs Standard Testing; Test type: Non-Inferiority — Self-testing was to be considered non-inferior with respect to the number of reported male CAI partners if the upper bound of the 95% CI for the fold-difference in the number of partners between the two arms (self ÷ standard testing) fell below 2; Poisson regression; [statistical method as in outcome 2, analysis 1]; Incidence Rate Ratio = 0.92, 95% CI 2-sided [0.64 to 1.33] — The home testing arm represents the numerator and the standard testing arm the denominator

ADVERSE EVENTS:
Time Frame: During study follow up (approximately 15 months)
Arm/Group | Home Testing | Standard Testing
Serious Adverse Events (participants affected / at risk) | 0/116 | 0/114
Other Adverse Events (participants affected / at risk) | 0/116 | 0/114

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes